CLINICAL TRIAL: NCT07080931
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Study on the Efficacy and Safety of 5% Minoxidil Foam in the Treatment of Female Androgenetic Alopecia
Brief Title: Efficacy and Safety of 5% Minoxidil Foam in Female Androgenetic Alopecia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang Sunshine Mandi Pharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-M2405(Foam)-lc
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Androgenetic Alopecia
Keywords: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5% Minoxidil Foam (Experimental)
  Interventions: Drug: 5% minoxidil foam
- Placebo for 5% Minoxidil Foam (Placebo Comparator)
  Interventions: Drug: Placebo for 5% Minoxidil Foam

INTERVENTIONS:
Drug: 5% minoxidil foam — Participants applied 5% minoxidil foam topically once daily (QD) in the morning or evening, with a maximum daily dose not exceeding 1 g, for up to 24 weeks.
  Arms: 5% Minoxidil Foam
Drug: Placebo for 5% Minoxidil Foam — Participants applied placebo once daily (QD) in the morning or evening, with a maximum daily dose not exceeding 1 g, for up to 24 weeks.
  Arms: Placebo for 5% Minoxidil Foam

SUMMARY:
The primary objective of this study is to evaluate the efficacy of once-daily 5% minoxidil foam versus placebo in female androgenetic alopecia, using the Target Area Terminal Hair Count (TAHC) as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the study and be able to provide a written Informed Consent Form (ICF);
* Female aged ≥ 18 years;
* Investigator-diagnosed androgenetic alopecia;
* Hair loss severity graded D3 to D6 on the Savin scale;
* Willingness to maintain identical hairstyle, hair color, and hair length at each follow-up visit;
* No pregnancy plans during the study and for 3 months post-last dose, with commitment to highly effective contraception. Women of childbearing potential must have negative serum pregnancy test ≤7 days prior to first investigational product administration

Exclusion Criteria:

* Study participants with known hypersensitivity to minoxidil or any excipient of the investigational product.
* Study participants with known hair loss disorders other than androgenetic alopecia (AGA)
* Study participants with any scalp disorder at screening that may interfere with efficacy evaluation, as determined by the investigator.
* Lactating women
* Study participants with history of hypotension or uncontrolled hypertension
* Study participants with clinically significant abnormal laboratory findings at screening that may compromise efficacy and safety assessments, as determined by the investigator.
* Study participants with clinically significant ECG abnormalities at screening
* Study participants with history of malignancy prior to screening.
* Study participants known to have conditions or disorders that may affect hair growth or compromise study results.
* Study participants with history of using systemically administered therapeutic drugs prior to screening that may interfere with efficacy evaluation, etc.
* Study participants with history of topical minoxidil application to alopecia-affected areas prior to screening.
* Study participants with no response to prior minoxidil treatment for alopecia
* Study participants with history of 5α-reductase inhibitor use prior to screening.
* Study participants with history of spironolactone or cyproterone treatment prior to screening.
* Study participants with history of autologous platelet-rich plasma (PRP) administration prior to screening.
* Study participants with history of chemotherapy, cytotoxic agents, scalp radiation, and/or low-level laser therapy (LLLT) or surgical scalp procedures for FAGA prior to screening.
* Study participants with history of using medical shampoos or solutions containing ingredients or other components that may interfere with efficacy evaluation prior to screening.
* Study participants planning hair transplantation during the study period, or using hair weaving, non-breathable wigs, or hair bonding during treatment.
* Study participants in other interventional clinical trials within 3 months before screening (excluding non-interventional studies and screen failures) , or planned concurrent clinical trial enrollment.
* Study participants with history of major surgery within 3 months before screening or planning major surgery during the study period.
* Study participants deemed by the investigator to have other conditions that may compromise compliance or render them unsuitable for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Target Area Hair Count (TAHC) at Week 24, assessed via digital phototrichogram analysis in study participa | Week 24

SECONDARY OUTCOMES:
Mean change from baseline in Target Area Hair Count (TAHC) at Weeks 6, 12, and 18 | Weeks 6, 12, and 18
Percent change from baseline in Target Area Hair Count (TAHC) at Weeks 12 and 24 | Weeks 12 , 24
Self-assessed satisfaction scores at Weeks 6, 12, 18, and 24 | Weeks 6, 12, 18, 24

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing, China, Beijing, China